CLINICAL TRIAL: NCT07126457
Title: A Randomized Controlled Study on the Improvement of Medical Experience for Patients With Radiation-induced Oropharyngeal Mucositis Based on the RIS System of the Internet of Things
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NFEC-2025-231
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer; Radiation-Induced Mucositis
Keywords: Radiation oropharyngeal mucositis; Head and Neck Cancer; Internet of things
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Use the RIS system
  Interventions: Other: RIS system
- control group (No Intervention): Do not use the ris system

INTERVENTIONS:
Other: RIS system — The RIS system based on the Internet of Things consists of three aspects: one-way output management of the large database of head and neck tumors, two-way interaction management of artificial intelligence applications, and popular science dissemination for the general public.
  Arms: experimental group

SUMMARY:
This study is a researcher-initiated, multi-center, prospective, two-arm interventional randomized controlled study across the country. It aims to explore whether an Internet of Things-based RIS system can enhance the medical experience of patients with radiation-induced oropharyngeal mucositis during the diagnosis and treatment process among head and neck cancer patients undergoing radiotherapy.

DETAILED DESCRIPTION:
After signing the informed consent form, patients who meet the inclusion/exclusion criteria will be randomly assigned in a 1:1 ratio to the experimental group (using the RIS system group) and the control group (not using the RIS system group), with a total of 110 patients recruited.

Subjects randomized to the experimental group will be managed and followed up using the RIS system based on Internet of Things technology from the start of radiotherapy until one year after radiotherapy.

Subjects randomized to the control group will be treated and followed up using the current clinical routine management model.

The treatment period refers to the time from the start of radiotherapy to one month after the end of radiotherapy. During this period, patients are treated according to the standard treatment methods for head and neck malignancies (concurrent chemoradiotherapy, induction chemotherapy followed by concurrent chemoradiotherapy, or radiotherapy alone, chemotherapy alone). In the experimental group, the RIS system is used for auxiliary management. After the start of radiotherapy, the three modules of the system (one-way output module, two-way interaction module, and public science popularization module) are used to manage patients until the end of the treatment period. The one-way output module management mainly transmits information to patients through the database, providing them with relevant suggestions such as precautions and psychological counseling. The two-way interaction module management mainly conducts interactive information exchange through artificial intelligence programs, providing patients with personalized and real-time life advice or precautions. The public science popularization module conducts science popularization education for the public and patients through popular science works.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form;
2. Reached the age of 18 on the date of signing the informed consent form, and under the age of 65;
3. Patients diagnosed with head and neck tumors and receiving radiotherapy as per the 2017 WHO standards and guidelines.
4. According to the doctor's assessment, patients may experience radiation-induced oropharyngeal mucositis during radiotherapy.

Exclusion Criteria:

* Have other uncontrolled serious diseases, such as unstable heart diseases requiring treatment, poorly controlled diabetes (fasting blood sugar > 1.5 times the upper limit of the normal value), mental disorders, and a severe history of allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
the satisfaction of patients | Through study completion, up to 3 years
  We use the patient satisfaction scale designed by us for the information age to assess patients' satisfaction during the diagnosis and treatment period.

SECONDARY OUTCOMES:
The response rate of the processing | Through study completion, up to 3 years
  The proportion of questions raised by the patients that were answered
Evaluation of response validity | Through study completion, up to 3 years
  The effectiveness score of the responses received to the patient's questions
The compliance rate of patients following the recommendations | Through study completion, up to 3 years
  The proportion of patients who followed the response advice and actually carried out the suggested actions
Doctor satisfaction | Through study completion, up to 3 years
  The satisfaction of doctors in the patient management process

CONTACTS AND LOCATIONS:
Overall Officials: Jian Guan, M.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (4):
- China (4):
  - Nanfang hospital, Southern medical university, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Jieyang people's hospital, Jieyang, Guangdong
  - Meizhou People's Hospital, Meizhou Academy of Medical Sciences Meizhou, Meizhou, Guangdong

IPD SHARING:
Plan to Share IPD: No